CLINICAL TRIAL: NCT06610422
Title: Association Between Neuropathy and Some Autoantibodies in Systemic Lupus Erythematosus (SLE) Patients With Lupus Nephritis in Assiut University Hospital
Brief Title: Association Between Neuropathy and Some Autoantibodies in Systemic Lupus Erythematosus (SLE) Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marina Asaad Fahmy Sedhom, Physician, Assiut University
Other Study IDs: Nephropathy and systemic lupus
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inactive stage: patients diagnosed as SLE and lupus nephritis (inactive stage)
- Active stage: patients diagnosed as SLE and lupus nephritis (active stage)
- Control: patients control group not SLE

SUMMARY:
1. Frequency of peripheral neuropathy associated with lupus nephritis
2. Sensitivity and specificity of some biomarkers used in diagnosis and follow up of SLE with lupus nephritis and peripheral neuropathy

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic, inflammatory,autoimmune disease that is characterized by multisystemic involvement with diverse clinical presentation .

Peripheral neuropathy is a well-documented clinical manifestation of systemic lupus erythematosus (SLE) , with a prevalence rate ranging from 2% to 27.8% . Several lines of evidence link the risk of neuropathy with the antiphospholipid antibody and rheumatoid factor , as well as neuropsychiatric lupus with anti-Ro . Some evidence links anti-ganglioside antibodies with neuropathy , but other studies do not . Peripheral neuropathy may be slowly progressive or acutely devastating . Lupus nephritis (LN), a more definite and specific subgroup of lupus, is a major cause of morbidity and mortality in SLE and can affect up to 60% of SLE patients. Furthermore, the presence of peripheral neuropathy in LN patients may be relevant for improving their lives . Such complex situation poses a therapeutic challenge. The clinical presentation of PN relies upon the diameter of the affected nerve, the sort of demyelinating or axonal lesions, and their acute or chronic occurrence . Routine nerve conduction studies just mirror the activity of the fast conducting myelinated A nerve fibers, which are physiologically irrelevant to pain. Hence, quantitative sensory testing can evaluate small nerve fiber function The pathogenesis of SLE-related neuropathy is obscure, and the few pathological studies of the peripheral nerves in SLE have revealed axonal degeneration, inflammatory changes, and vasculitis .

The major inflammatory mediators released from immune cells act on sensory neurons, inducing peripheral sensitization and hyperalgesic phenomena. In addition, after damage, this natural inflammatory response could encourage the pathogenetic activity of antineural autoantibodies, in addition to ischemic vascular mechanism, by vasa nervorum vascularitis or by microthrombi linked to antiphospholipid antibodies.

The other legitimate mechanisms are immunologic cause by a direct aggression by antibodies, entraining obliteration of the peripheral nerve component.

Furthermore, the PN has not been well prescribed in SLE in terms of onset, severity, clinical associations, and electrophysiological characteristics.. Therefore, we are going to characterize PN in SLE with respect to the patient's clinical lupus properties, serologic markers, disease activity, and electrophysiological data

ELIGIBILITY:
Inclusion Criteria:

* 1. Female patients

  2. Age ≥ 18 years

  3. Patients diagnosed as SLE and lupus nephritis as clinical, laboratory investigations and renal biopsy for indicated cases 4. Anti phospholipid antibodies (IgG & IgM) 5.Associated vasculitis ( cANCA & pANCA ) 6.Active - inactive classes of SLE 7.CKD stage I & IV not on dialysis

Exclusion Criteria:

* 1.history of viral hepatitis B or C 2.A history of malignancy (excluding basal cell carcinoma) 3.pulse therapy 4.chronic kidney disease (CKD) stage 5 or hemodialysis 5.SLE not associated with renal affect

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, ):patients demographics including )age ,sex , residence , occupation,age at time of diagnosis) Full history and examination
  Laboratory data & Investigations
  1. CBC
  2. Kidney function tests
  3. ESR
  4. CRP
  5. urine analysis
  6. screening for (HBv- HcV-HIV)
  7. Autoantibodies: ANA , Anti- ds DNA
  8. Rheumatoid factor
  9. neuromuscular ultrasound 10 - nerve conduction
Sampling Method: Non-Probability Sample
Enrollment: 159 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Nephropathy and autoantibodies | through study completion, an average of 1 year]]
  1- Relation between neuropathy and autoantibodies in lupus nephritis
Prepherial nephropathy and systemic lupus | through study completion, an average of 1 year]
  Evaluate the frequency and severity of symptoms of peripheral neuropathy among patients with lupus nephritis
Electrophysiology | through study completion, an average of 1 year]]
  Study electrophysiological properties of peripheral neuropathy and their relation to disease activity